CLINICAL TRIAL: NCT06253286
Title: Predictability of Part-time Wearing of Removable Clear Aligner Therapy Versus Full Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Mohamed Adel Zein, Principle Investigator, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUE.REC (24)/11-2020
Record Dates: First submitted 2021-06-27; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Malocclusion, Angle Class I
MeSH Terms: conditions — Malocclusion, Angle Class I

STUDY DESIGN:
Intervention Model Description: A randomized controlled clinical trial of 2 parallel groups with an allocation ratio of 1:1
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- part-time wear (Active Comparator): Patients will be instructed to wear the aligner for 16 hours per day, then the aligner going to be changed to the next step according to its numerical order in the software
  Interventions: Device: clear aligner treatment for orthodontics patients
- Full-time wear (Active Comparator): Patients will be instructed to wear the aligner for 22 hours per day, then the aligner going to be changed to the next step according to its numerical order in the software
  Interventions: Device: clear aligner treatment for orthodontics patients

INTERVENTIONS:
Device: clear aligner treatment for orthodontics patients — patient are instructed to wear aligners

SUMMARY:
14 Patients with mild to moderate crowding and spacing will be selected according to inclusion criteria.

Treatment planning will be done on Maestro® software. An impression will be taken and scanned by an extra-oral scanner. The models will be 3D printed and aligner trays will be fabricated to be delivered on biweekly basis to be worn 16 hours per day for one group and 22 hours for the other group. Superimposition of the achieved clinical model over the predicted model will be done. Linear and angular measurements will be calculated for each tooth.

DETAILED DESCRIPTION:
Clear removable retainers could be related to clear aligners. Wearing time of retainers has been suggested that it could be changed from full time to part-time during the night only. A similar approach could be done to determine the effect of wearing time of clear aligners on treatment outcome. The standard duration per day for wearing the appliance is 22 hours. However, is part-time wearing (16 hours) would have the same effect? Therefore, a randomized clinical trial is needed to compare the effect of partial wearing of the aligner versus full time. Moreover, studying the predictability and accuracy of treatment using Maestro software.

ELIGIBILITY:
Inclusion Criteria:

1. Permeant dentition
2. Mild to moderate crowding and spacing in maxilla and mandible according to Little's Irregularity Index
3. Non-extraction cases

Exclusion Criteria:

1. Severe crowding and spacing
2. Systematic diseases
3. Compromised periodontal health
4. Craniofacial syndromes

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Linear Movement Discrepancies Between Digital Software Models and Clinical Models | an average of 1 year
  Translation movements (mm) were compared for each tooth between predicted models on Software predicted models and actual clinical models for the study groups
Angular Movement Discrepancies Between Digital Software Models and Clinical Models | an average of 1 year
  Translation movements (Degrees) were compared for each tooth between predicted models on Software predicted models and actual clinical models for the study groups

CONTACTS AND LOCATIONS:
Overall Officials: Hala Mounir, Prof, Study Chair — Future University in Egypt
Locations (1):
- Future University in Egypt, Cairo, New Caro, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The trial results will be available to the participants, health care professionals and the public by publication of the study in high quality national and international journals. The principal investigator will present a copy of the thesis at the Faculty of Oral and Dental Medicine, Future University in Egypt library and will distribute additional copies among the main universities in Egypt.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after publication, indefinitely
Access Criteria: Professors of other institutions will have access to the data if required via email

REFERENCES:
- [Background] Nahoum HI. Forces and moments generated by removable thermoplastic aligners. Am J Orthod Dentofacial Orthop. 2014 Nov;146(5):545-6. doi: 10.1016/j.ajodo.2014.08.006. Epub 2014 Oct 28. No abstract available. PMID 25439196
- [Background] Djeu G, Shelton C, Maganzini A. Outcome assessment of Invisalign and traditional orthodontic treatment compared with the American Board of Orthodontics objective grading system. Am J Orthod Dentofacial Orthop. 2005 Sep;128(3):292-8; discussion 298. doi: 10.1016/j.ajodo.2005.06.002. PMID 16168325
- [Background] Papadimitriou A, Mousoulea S, Gkantidis N, Kloukos D. Clinical effectiveness of Invisalign(R) orthodontic treatment: a systematic review. Prog Orthod. 2018 Sep 28;19(1):37. doi: 10.1186/s40510-018-0235-z. PMID 30264270
- [Background] Melsen B. Northcroft lecture: how has the spectrum of orthodontics changed over the past decades? J Orthod. 2011 Jun;38(2):134-43; quiz 145. doi: 10.1179/14653121141362. PMID 21677105
- [Background] Pratt MC, Kluemper GT, Lindstrom AF. Patient compliance with orthodontic retainers in the postretention phase. Am J Orthod Dentofacial Orthop. 2011 Aug;140(2):196-201. doi: 10.1016/j.ajodo.2010.02.035. PMID 21803257
- [Background] Kacer KA, Valiathan M, Narendran S, Hans MG. Retainer wear and compliance in the first 2 years after active orthodontic treatment. Am J Orthod Dentofacial Orthop. 2010 Nov;138(5):592-8. doi: 10.1016/j.ajodo.2008.12.027. PMID 21055599
- [Background] Jacox LA, Mihas P, Cho C, Lin FC, Ko CC. Understanding technology adoption by orthodontists: A qualitative study. Am J Orthod Dentofacial Orthop. 2019 Mar;155(3):432-442. doi: 10.1016/j.ajodo.2018.08.018. PMID 30826046
- [Background] Alford TJ, Roberts WE, Hartsfield JK Jr, Eckert GJ, Snyder RJ. Clinical outcomes for patients finished with the SureSmile method compared with conventional fixed orthodontic therapy. Angle Orthod. 2011 May;81(3):383-8. doi: 10.2319/071810-413.1. Epub 2011 Jan 24. PMID 21261488
- [Background] Brown MW, Koroluk L, Ko CC, Zhang K, Chen M, Nguyen T. Effectiveness and efficiency of a CAD/CAM orthodontic bracket system. Am J Orthod Dentofacial Orthop. 2015 Dec;148(6):1067-74. doi: 10.1016/j.ajodo.2015.07.029. PMID 26672713
- [Background] Kravitz ND, Kusnoto B, BeGole E, Obrez A, Agran B. How well does Invisalign work? A prospective clinical study evaluating the efficacy of tooth movement with Invisalign. Am J Orthod Dentofacial Orthop. 2009 Jan;135(1):27-35. doi: 10.1016/j.ajodo.2007.05.018. PMID 19121497
- [Background] Zhang XJ, He L, Guo HM, Tian J, Bai YX, Li S. Integrated three-dimensional digital assessment of accuracy of anterior tooth movement using clear aligners. Korean J Orthod. 2015 Nov;45(6):275-81. doi: 10.4041/kjod.2015.45.6.275. Epub 2015 Nov 20. PMID 26629473
- [Background] Buschang PH, Ross M, Shaw SG, Crosby D, Campbell PM. Predicted and actual end-of-treatment occlusion produced with aligner therapy. Angle Orthod. 2015 Sep;85(5):723-7. doi: 10.2319/043014-311.1. Epub 2014 Nov 5. PMID 25372019
- [Background] Weir T. Clear aligners in orthodontic treatment. Aust Dent J. 2017 Mar;62 Suppl 1:58-62. doi: 10.1111/adj.12480. PMID 28297094
- [Background] Grunheid T, Loh C, Larson BE. How accurate is Invisalign in nonextraction cases? Are predicted tooth positions achieved? Angle Orthod. 2017 Nov;87(6):809-815. doi: 10.2319/022717-147.1. Epub 2017 Jul 7. PMID 28686090
- [Background] Rossini G, Parrini S, Castroflorio T, Deregibus A, Debernardi CL. Efficacy of clear aligners in controlling orthodontic tooth movement: a systematic review. Angle Orthod. 2015 Sep;85(5):881-9. doi: 10.2319/061614-436.1. Epub 2014 Nov 20. PMID 25412265
- [Background] Simon M, Keilig L, Schwarze J, Jung BA, Bourauel C. Treatment outcome and efficacy of an aligner technique--regarding incisor torque, premolar derotation and molar distalization. BMC Oral Health. 2014 Jun 11;14:68. doi: 10.1186/1472-6831-14-68. PMID 24923279
- [Background] Charalampakis O, Iliadi A, Ueno H, Oliver DR, Kim KB. Accuracy of clear aligners: A retrospective study of patients who needed refinement. Am J Orthod Dentofacial Orthop. 2018 Jul;154(1):47-54. doi: 10.1016/j.ajodo.2017.11.028. PMID 29957318
- [Background] Izhar A, Singh G, Goyal V, Singh R, Gupta N, Pahuja P. Comparative Assessment of Clinical and Predicted Treatment Outcomes of Clear Aligner Treatment: An in Vivo Study. Turk J Orthod. 2019 Dec 1;32(4):229-235. doi: 10.5152/TurkJOrthod.2019.19019. eCollection 2019 Dec. PMID 32110468
- [Background] Lombardo L, Arreghini A, Ramina F, Huanca Ghislanzoni LT, Siciliani G. Predictability of orthodontic movement with orthodontic aligners: a retrospective study. Prog Orthod. 2017 Nov 13;18(1):35. doi: 10.1186/s40510-017-0190-0. PMID 29130127
- [Background] Chisari JR, McGorray SP, Nair M, Wheeler TT. Variables affecting orthodontic tooth movement with clear aligners. Am J Orthod Dentofacial Orthop. 2014 Apr;145(4 Suppl):S82-91. doi: 10.1016/j.ajodo.2013.10.022. PMID 24680028
- [Background] Thickett E, Power S. A randomized clinical trial of thermoplastic retainer wear. Eur J Orthod. 2010 Feb;32(1):1-5. doi: 10.1093/ejo/cjp061. Epub 2009 Oct 14. PMID 19828592
- [Background] Gill DS, Naini FB, Jones A, Tredwin CJ. Part-time versus full-time retainer wear following fixed appliance therapy: a randomized prospective controlled trial. World J Orthod. 2007 Fall;8(3):300-6. PMID 17902334
- Available data/document: Study Protocol — https://drive.google.com/file/d/1edivKccFOAyt3_A6aNnNROe7JQnRmp4C/view?usp=sharing
- Available data/document: Informed Consent Form — https://drive.google.com/file/d/1gA2nThyz6di3bSZKJQ7aQ_Usy1_wpOrR/view?usp=sharing